CLINICAL TRIAL: NCT03644290
Title: Neural Correlates and Functional Connectivity Associated With Cognitive Memory Training in Patients With Cerebral Ischemic Lesions
Brief Title: Cognitive Training in Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: São Paulo State University (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Eliane Mioto, Principal investigator, São Paulo State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Stroke Rehab
Record Dates: First submitted 2018-08-16; First posted 2018-08-23 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Vascular Diseases
Keywords: vascular ischemic lesion
MeSH Terms: conditions — Vascular Diseases | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive training (Experimental): Semantic categorization training sessions
  Interventions: Behavioral: Cognitive training
- Control condition (Active Comparator): Five sessions of behavioral control condition with information and education
  Interventions: Behavioral: Control Condition

INTERVENTIONS:
Behavioral: Cognitive training — Five sessions of semantic strategy training and face-name association training
  Arms: Cognitive training
Behavioral: Control Condition — Five sessions of active control information and education
  Arms: Control condition

SUMMARY:
The study aims to investigate the behavioral effects, neural correlates and functional connectivity of cognitive training in patients with stroke

DETAILED DESCRIPTION:
The study will investigate the effects of two cognitive training strategies on behavior, neural correlates and functional connectivity of patients with vascular lesions. The first strategy is associated to the ability to apply efficient organizational semantic category strategy to a list of words. This strategy will be trained in activities similar to everyday life activities. There will be in total 5 sessions, two for measuring the generalization effects before and after training and three sessions to apply the semantic strategy in order to improve encoding and episodic memory performance. The second strategy is related to the ability to remember face-names and the strategy will involve the identification of a salient face feature, creation of a nickname and association of the nickname to the real name. There will be 5 sessions in total, two for measuring the generalization effects before and after training and three sessions to apply the face-name association strategy in order to improve encoding and episodic memory performance. These two cognitive training procedures will be carried out in two separate moments. Before and after each procedure all participants will be examined by functional MRI during resting state and during a active task using a memory encoding paradigm. The same procedure will be carried out with normal control participants.

ELIGIBILITY:
Inclusion Criteria:

* people with chronic vascular ischemic lesions (more than 6 months)

Exclusion Criteria:

* vascular hemorrhages, stenosis, psychiatric problems

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-01-02 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline memory performance at 6 months | up to 24 weeks after intervention
  Hopkins Verbal Learning Test (episodic memory test total immediate score 48 and delayed score12) and fMRI active task (news recall immediate and delayed score 12)

SECONDARY OUTCOMES:
Change from baseline everyday life activity performance at 6 months | up to 24 weeks of intervention
  Generalization questionnaire (questions on difficulties in everyday memory total score 12)

CONTACTS AND LOCATIONS:
Overall Officials: Eliane C Miotto, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gibson E, Koh CL, Eames S, Bennett S, Scott AM, Hoffmann TC. Occupational therapy for cognitive impairment in stroke patients. Cochrane Database Syst Rev. 2022 Mar 29;3(3):CD006430. doi: 10.1002/14651858.CD006430.pub3. PMID 35349186
- [Derived] Miotto EC, Bazan PR, Batista AX, Conforto AB, Figueiredo EG, Martin MDGM, Avolio IB, Amaro E Jr, Teixeira MJ. Behavioral and Neural Correlates of Cognitive Training and Transfer Effects in Stroke Patients. Front Neurol. 2020 Sep 15;11:1048. doi: 10.3389/fneur.2020.01048. eCollection 2020. PMID 33041987